CLINICAL TRIAL: NCT05677516
Title: Incidence and Duration of Unintentional Neuromodulation Effects After Pulmonary Vein Isolation in Patients With Atrial Fibrillation. (UNCOVER-PVI)
Brief Title: Incidence and Duration of Unintentional Neuromodulation Effects After Pulmonary Vein Isolation in Patients With Atrial Fibrillation.
Acronym: UNCOVER-PVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: 4th Military Clinical Hospital with Polyclinic, Poland (Other)
Responsible Party: Principal Investigator, Krystian Josiak, PhD, 4th Military Clinical Hospital with Polyclinic, Poland
Other Study IDs: UNCOVER-PVI
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Atrial Fibrillation
Keywords: pulmonary vains isolation, catdioneuroablation, cardioneuromodultion
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electrocardiography, Ambulatory; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Patients undergoing cryoablation of pulmonary veins with paroxysmal or persistent AF with ongoing AF during ablation.
  Interventions: Procedure: ablation- pulmonary vain isolation- crioablation; Procedure: Electrophysiological study (EPS); Diagnostic Test: Holter EKG; Other: Questionnaire
- Group 2: Patients undergoing cryoablation of pulmonary veins with paroxysmal AF, in sinus rhythm during the procedure.
  Interventions: Procedure: ablation- pulmonary vain isolation- crioablation; Procedure: Electrophysiological study (EPS); Diagnostic Test: Holter EKG; Other: Questionnaire
- Group 3: Patients undergoing pulmonary veins isolation with PFA with paroxysmal AF, in sinus rhythm during the procedure.
  Interventions: Procedure: ablation- pulmonary vain isolation- pulsed field ablation (PFA); Procedure: Electrophysiological study (EPS); Diagnostic Test: Holter EKG; Other: Questionnaire
- Group 4: Patients undergoing RF ablation of the pulmonary veins using an electroanatomical system with paroxysmal AF, in sinus rhythm during the procedure.
  Interventions: Procedure: ablation- pulmonary vain isolation- radiofrequency ablation (RF); Procedure: Electrophysiological study (EPS); Diagnostic Test: Holter EKG; Other: Questionnaire

INTERVENTIONS:
Procedure: ablation- pulmonary vain isolation- crioablation — Pulmonary vein isolation is the electrical isolation of the pulmonary veins from the left atrium. It can be performed using the cryoablation technique. The procedure begins with venous access through the femoral vein through which catheters and electrodes are inserted. Then, the left atrium is accessed through a transseptal puncture and the pulmonary veins are isolated using a cryoablation balloon. Cryoablation procedures are performed under local anesthesia. The procedure is performed using X-ray fluoroscopy.
  Groups: Group 1; Group 2
Procedure: ablation- pulmonary vain isolation- pulsed field ablation (PFA) — Pulmonary vein isolation is the electrical isolation of the pulmonary veins from the left atrium. It can be performed using the pulsed field ablation (PFA) technique. The procedure begins with venous access through the femoral vein through which catheters and electrodes are inserted. Then, the left atrium is accessed through a transseptal puncture and the pulmonary veins are isolated with a PFA electrode. PFA procedures are performed under general anesthesia. The procedure is performed using X-ray fluoroscopy.
  Groups: Group 3
Procedure: ablation- pulmonary vain isolation- radiofrequency ablation (RF) — Pulmonary vein isolation is the electrical isolation of the pulmonary veins from the left atrium. It can be performed using the radiofrequency ablation (RF) technique. The procedure begins with venous access through the femoral vein through which catheters and electrodes are inserted. Then, the left atrium is accessed through a transseptal puncture and the pulmonary veins are isolated with a RF electrode. RF procedures are performed under local anesthesia. The procedure is performed using X-ray fluoroscopy.
  Groups: Group 4
Procedure: Electrophysiological study (EPS) — In the electrophysiological study (EPS), electrophysiological parameters such as the recovery time of sinus rhythm (SNRT), Wenckebach's point, AH and HV intervals are measured. The examination begins with venous access through the femoral vein. Then, diagnostic electrodes are inserted into the right atrium, right ventricle and coronary sinus, with which electrophysiological tests are performed. The SNRT is measured after 60 seconds of atrial pacing with a 600ms cycle. The Wencjabach point is determined by stimulation in the incremental protocol. AV and HV intervals are measured during sinus rhythm using an electrode placed on the bundle of His. EPS is performed under local anesthesia. EPS will be performed both before and after pulmonary vein isolation. In patients with atrial fibrillation, during ablation, only the HV interval will be measured.
  The procedure is performed using X-ray fluoroscopy.
Diagnostic Test: Holter EKG — Holter ECG is a 24-hour, non-invasive ECG recording using a portable recorder and electrodes placed on the patient's chest. The Holter ECG will be performed three times: on the day preceding and on the first day after pulmonary veins isolation, and after 3 months of observation.
Other: Questionnaire — The survey will be conducted after 3 months of observation and will include questions about the number of hospitalizations due to atrial fibrillation, heart palpitations, changes in pharmacotherapy.

SUMMARY:
Pulmonary vein isolation (PVI) is a proven, high-efficiency treatment for atrial fibrillation (AF). Performed, among others, using cryoablation, pulsed field ablation (PFA) or radiofrequency (RF) ablation. It has been shown that its effectiveness significantly increases when the PVI procedure is combined with cardioneuroablation (CNA). The autonomic nervous system - ganglionated plexi (GP), the target of the CNA, are the endings of the vagal nerve and are located in the neighborhood of the pulmonary veins ostia. Places that, in many cases, are unintentionally damaged during PVI. Varying degrees of injury to the GP during PVI indicate that the group of patients undergoing PVI is heterogeneous in this regard, and the effectiveness of PVI may vary. Vagal nerve endings damage during CNA abolishes or modifies its activity, which is manifested by the acceleration of sinus rhythm and increased atrioventricular conduction efficiency. Unintended CNA is not observed in every PVI procedure. The severity of the unintended CNA effect and its duration also vary.

THE STUDY OBJECTIVES:

1. Frequency of unintentional CNA occurrence during PVI
2. Duration effect of CNA after unintentional CNA
3. Evaluation of the relationship between the different kinds of energy - cryo, pulsed field) and RFwith the unintentional CNA frequency occurrence and durability effect
4. Clinical significance evaluation of the new assessment method of the CNA effectiveness with the measure of the cSNRT and the sinus rate after its return, measured before and after PVI
5. Assessment of clinical significance for CNA evaluation of the electrophysiological parameters of AV node conduction efficiency, such as PQ interval, AH interval, HV interval, and Wenckebach's point. Parameters will be examined before and after PVI.
6. PVI efficacy evaluation with the AF and Sick Sinus Syndrome treatment, especially with the elimination of the indications for the PM implantation (sinus bradycardia, AV conduction disorders)
7. Assessment of sinus rhythm maintenance after PVI with unintentional CNA and without unintentional CNA
8. Assessment of ventricular rate control during AF burden after unintentional CNA
9. The search for new parameters evaluating the effectiveness and degree of CNA, such as the change in SR frequency after its return, may prove helpful and allow for resignation or significantly reduce the use of the complicated protocol of extracardiac vagal ganglion stimulation (ECVS) as a method to verify the effectiveness CNAs.

DETAILED DESCRIPTION:
This is a multi-centre, prospective, observational study, which will include patients with paroxysmal or persistent atrial fibrillation qualified for PVI by the European Society of Cardiology guidelines. Pulmonary veins will be isolated with three kinds of energies: cryo, pulsed field and RF. The study group will consist of four subgroups:

1. Patients undergoing cryoablation of pulmonary veins with paroxysmal or persistent AF with ongoing AF during ablation
2. Patients undergoing cryoablation of pulmonary veins with paroxysmal AF, in sinus rhythm during the procedure
3. Patients undergoing pulmonary veins isolation with PFA with paroxysmal AF, in sinus rhythm during the procedure
4. Patients undergoing RF ablation of the pulmonary veins using an electroanatomical system with paroxysmal AF, in sinus rhythm during the procedure

The effect of unintentional neuromodulation will be assessed based on the following:

1. ECG Holter monitoring performed before and after the procedure in all groups
2. Parameters assessed in EPS before and after the procedure in groups 2,3, and 4.

The long-term effect of neuromodulation and its impact on maintaining sinus rhythm will be assessed based on the following:

1. The Holter ECG monitoring in groups 2,3, and 4.
2. The interview in all groups after three months of observation.

PROTOCOL STUDY:

GROUP 1:

1. Holter ECG prior to PVI
2. Holter ECG after PVI
3. Survey after three months of observation.

GROUPS 2,3 AND 4:

1. Holter ECG prior to PVI
2. EPS prior to PVI
3. EPS after PVI
4. Holter ECG prior to PVI
5. Holter ECG after three to six months of observation
6. Survey after three months of observation.

All the measured parameters as well as demographic and clinical data will be recorded in the study database.

ELIGIBILITY:
Inclusion Criteria:

* Patients qualified for PVI due to paroxysmal or persistent atrial fibrillation.
* Signed and dated written informed consent prior to admission to the trial.

Exclusion Criteria:

* Any underwent cardiac ablation.
* A history of cardiac surgery.
* Pregnancy.
* Diseases affecting the autonomic nervous system.
* Change in heart rhythm during PVI, with no conversion to the primary rhythm at the end of the procedure.
* Cardiac pacing during Holter ECG monitoring.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group will consist of patients aged 18-85. With paroxysmal or persistent atrial fibrillation. Qualified for PVI according to the guidelines of the European Society of Cardiology.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-12-23 (Estimated); Study Completion 2023-12-23 (Estimated)

PRIMARY OUTCOMES:
Acceleration and maintenance of a faster sinus rhythm after PVI | 3 months of follow-up
  Based on EPS before and after PVI and Holter ECG before and after PVI and after 3 months of follow-up.
Improvement of AV conduction efficiency and its durability after PVI | 3 months of follow-up
  Based on EPS before and after PVI and Holter ECG before and after PVI and after 3 months of follow-up.
Recurrence of AF during the observation period. | 3 months of follow-up
  Based on Holter ECG and survey after 3 months of follow-up.

SECONDARY OUTCOMES:
AF recurrence with the need to increase doses of heart rate control drugs. | 3 months of follow-up
  Based on survey after 3 months of follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - 4th Military Hospital, Cardiology Department, Wroclaw, Lower Silesian Voivodeship
  - Polish-American Heart Clinics Cardiovascular Center in Dąbrowa Górnicza, American Heart of Poland Group, Dąbrowa Górnicza, Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: No
The data will be collected in a database accessible only to the named researchers.

REFERENCES:
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Katritsis DG, Pokushalov E, Romanov A, Giazitzoglou E, Siontis GC, Po SS, Camm AJ, Ioannidis JP. Autonomic denervation added to pulmonary vein isolation for paroxysmal atrial fibrillation: a randomized clinical trial. J Am Coll Cardiol. 2013 Dec 17;62(24):2318-25. doi: 10.1016/j.jacc.2013.06.053. Epub 2013 Aug 21. PMID 23973694
- [Background] Aksu T, Guler TE, Bozyel S, Yalin K, Gopinathannair R. Why is pulmonary vein isolation not enough for vagal denervation in all cases? Pacing Clin Electrophysiol. 2020 May;43(5):520-523. doi: 10.1111/pace.13922. Epub 2020 May 2. PMID 32324285
- [Background] Sakamoto S, Schuessler RB, Lee AM, Aziz A, Lall SC, Damiano RJ Jr. Vagal denervation and reinnervation after ablation of ganglionated plexi. J Thorac Cardiovasc Surg. 2010 Feb;139(2):444-52. doi: 10.1016/j.jtcvs.2009.04.056. Epub 2009 Sep 9. PMID 19740492
- [Background] Yorgun H, Aytemir K, Canpolat U, Sahiner L, Kaya EB, Oto A. Additional benefit of cryoballoon-based atrial fibrillation ablation beyond pulmonary vein isolation: modification of ganglionated plexi. Europace. 2014 May;16(5):645-51. doi: 10.1093/europace/eut240. Epub 2013 Aug 16. PMID 23954919